CLINICAL TRIAL: NCT02400203
Title: FREE Living Hulled HEMP Seed and Oil Trial
Acronym: FREEHEMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B2014:115-2
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Overweight
Keywords: hemp oil,; hemp; fatty acids; omega-6; omega-3; blood pressure; blood lipids
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): 54 grams of hulled sesame seeds, consumed in 2 daily 27 gram portions, and 30 grams of soybean oil per day
  Interventions: Other: Control
- Hemp foods (Experimental): 60 grams of hulled hemp seeds,consumed in 2 daily 30 gram portions, and 30 grams of hemp oil per day
  Interventions: Other: Hemp foods

INTERVENTIONS:
Other: Control
  Arms: Control
Other: Hemp foods
  Arms: Hemp foods

SUMMARY:
The objectives of this trial are to assess the effects of hemp product consumption, specifically hulled hemp seeds and hemp oil on blood fatty acid profiles and cardiovascular disease risk factors, in healthy overweight volunteers after 4 weeks of consumption.

DETAILED DESCRIPTION:
The trial will be a 4 week double-blinded, randomized, cross-over design with 2 treatment intervention (hemp and control) periods separated by a 4 week washout period. Thirty metabolically healthy overweight volunteers will be recruited into the trial.

On day 1, and 27, 28 of each treatment period participants will be asked to come to the Richardson Center for Functional Foods and Nutraceuticals (RCFFN) for a 12 hour fasted blood sample. On day 1, participants will be given prepackaged sachets of treatment hulled seeds (hemp or sesame) and salad dressing, containing 30 g/d of treatment (hemp or soybean) oil (in individually packaged daily containers) will also be supplied.

Participants will be instructed by clinical coordinators to integrate the products (2 sachets of seeds, 1 salad dressing) into their daily meals and to avoid other dietary sources of n-3 fatty acids, such as flax, chia, camelina, krill and fish products. Participants will be given activity monitors to wear during the intervention periods. Participants will be required to eat one sachet of hulled seeds in the morning and one in the evening, and to consume the dressing throughout the day, for each 4 week treatment period.

Participants will be asked to continue their habitual diets, while avoiding large dietary sources of n-3 fatty acids, throughout the treatment and washout periods. Participants will be instructed to maintain the same level of physical activity and alcohol intake throughout the trial period. The trial coordinator will contact participants weekly via telephone or email to monitor treatment adherence and to answer any questions or concerns participants might have. Background dietary intakes will be measured at day 1 of the trial using a food frequency questionnaire, and during each treatment period by 3-day food record to be completed in the last week of each treatment period. Participants will be asked questions about the interventions including side effects, mood and perceived energy level by trial coordinators at the end of each intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Metabolically healthy overweight (BMI 25-35 kg/m2) participants aged 18-65,
* Men and women with the ability to give written informed consent and comply with trial guidelines.

Exclusion Criteria:

* Pregnancy or lactation
* Smokers (tobacco products for the last 6 months)
* History of cancer, rheumatoid arthritis, chronic illness, cardiovascular problems, liver and kidney disease, inflammatory bowel disease, pancreatitis, gallbladder or biliary disease, neurological/psychological disease, bleeding disorders, experienced platelet abnormalities, and gastrointestinal disorders that could interfere with fat absorption, serum glucose over ≥6.1 mmol/L, serum triglycerides (TG) >4.52 mmol/L, and/or LDL cholesterol (LDL-C) ≥6.5 mmol/L, hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg),
* Body mass index (BMI; in kg/m2) ≥35
* Consume or plan to consume anticoagulant,
* Hypertension or lipid lowering medications, or hypotensive
* Lipid lowering or n-3 PUFA dietary supplements
* Reported consumption of more than 2 alcoholic drinks/day or history of alcoholism or drug dependence
* Reported use of any experimental medication within 1 month prior to starting the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change in red blood cell omega-3 fatty acid content | Baseline (Day 1) and Endpoint (Day 27,28) of each experimental period
  Total lipids will be extracted from each fraction (whole plasma, RBC) and will be evaluated for its fatty acid composition using gas-chromatography linked with flame ionization detector

SECONDARY OUTCOMES:
Change in plasma lipids | Baseline (Day 1) and Endpoint (Day 27,28) of each experimental period
  TC, HDL-C and TG in serum, will be determined by automated methods in duplicate on an auto-analyzer (VITROS 350). LDL-C concentrations will be calculated using the Friedewald equation.
Change in inflammatory and endothelial function biomarkers | Baseline (Day 1) and Endpoint (Day 27,28) of each experimental period
  Measurement of inflammatory biomarker such as CRP, IL-6 and TNF-α and cell adhesion molecules such as e-selectin, p-selectin, s-ICAM and s-VCAM, will be measured in multiplex on a Meso Scale Discovery platform.
Change in blood pressure and arterial stiffness | Baseline (Day 1) and Endpoint (Day 27,28) of each experimental period
  Blood pressure will be measure in conjunction with pulse wave velocity (PWV) and augmentation index (AI) to assess arterial stiffness using a Mobil-O-Graph, in triplicate.
Change in glucose metabolism and insulin sensitivity | Baseline (Day 1) and Endpoint (Day 27,28) of each experimental period
  Measurement of fasting glucose using an auto-analyzer, and insulin by radioimmunoassay, to investigate the impact of hemp product consumption on glucose metabolism and insulin sensitivity.

OTHER OUTCOMES:
Change in body composition | Measurements will be done at the beginning and end of each of the two 4-week treatment
  Using a Dual Energy X-Ray Absorptiometry machine to analyze body composition, including measuring visceral adiposity
Physical activity | from day 20-28 of each treatment period
  The activity monitors will measure the participants' physical activity levels, steps taken, and the different amounts of time spent at different activity levels.

CONTACTS AND LOCATIONS:
Overall Officials: Rotimi Aluko, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba, Canada